CLINICAL TRIAL: NCT07406425
Title: Evaluation of Efficacy of Coconut Oil Mouth Care for Non-autonomous Hospitalised Elderly People: a Multicentric Randomised Controlled Trial
Brief Title: Evaluation of Efficacy of Coconut Oil Mouth Care for Non-autonomous Hospitalised Elderly People.
Acronym: COCO-CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 87RI24_0064 (COCO-CARE)
Record Dates: First submitted 2026-01-20; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Geriatrics; Oral Health Care
Keywords: geriatrics; oral health care; elderly; coconut oil; palliative care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coconut oil mouth care (Experimental): Daily oral care is done with coconut oil throughout the patient's hospitalization
  Interventions: Procedure: Coconut oil mouth care
- Glycerin mouthwashes (Active Comparator): Daily oral care is performed with glycerin sticks as in current practice.
  Interventions: Procedure: Glycerin mouthwashes

INTERVENTIONS:
Procedure: Coconut oil mouth care — Daily oral care is done with coconut oil throughout the patient's hospitalization
  Arms: Coconut oil mouth care
Procedure: Glycerin mouthwashes — Daily oral care is performed with glycerin sticks as in current practice.
  Arms: Glycerin mouthwashes

SUMMARY:
This is a prospective, longitudinal, randomised, open-label, multicentric, interventional, comparative superiority study.

The main objective is to demonstrate the superiority of oral care with coconut oil on the oral status of elderly people hospitalised in geriatrics, versus oral care with glycerol sticks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 and over
* Patients hospitalised in geriatric medicine and geriatric SMR departments
* Patients able to open their mouths for treatment
* Patients not able to carry out their oral hygiene on their own
* Patients who have given their written consent (consent of the patient or patient consent accompanied by the designated representative if the patient is unable to give written consent)

Exclusion Criteria:

* Patients with a known allergy to coconut
* Patients requiring medicated mouth care as prescribed by a doctor
* Patients under guardianship, tutorship or curatorship
* Confused patients who have had medically diagnosed dehydration for less than 48 hours
* Patients with swallowing difficulties
* Patients in the terminal phase of end of life

Secondary exclusion criteria:

* Patients leaving the department between D1 and D8 (whatever the reason for discharge, and including in the event of death)
* Patients whose condition progresses towards a terminal phase of the end of life between D1 and D8
* Patients experiencing an allergic reaction to Coconut Oil during the study
* Patients who may present with dehydration during the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Revised Oral Assement Guide (ROAG) between Day 1 and Day 8 | From Day 1 to Day 8
  Change in total score between Day 1 (D1) and Day 8 (D8) on the Revised Oral Assessment Guide (ROAG), translated and validated in French.
  The scale assesses 8 indicators (voice, swallowing, lips, tongue,saliva, mucous membranes, gums and teeth) according to 3 levels. The result gives a total score out of 24 points

SECONDARY OUTCOMES:
Weekly ROAG scores (Revised Oral Assment Guide) | Every week from the date of inclusion until the date of discharge, on average over 37 days.
  Weekly ROAG scores (overall score and score per indicator) for all participants included until discharge (an assessment will also be carried out at discharge).
ROAG betwen Day 1 (D1) and Day 8 (D8) for patients with "palliative care" status | from Day 1 to Day 8
  Changes in the ROAG overall score between D1 and D8, translated and validated in French. The degree of dependence is assessed using the KATZ scale (dependence group) at inclusion.
Number of oral care stopped | At the end of the study, on average of 37 days.
  Number of patients who stopped the oral care initially proposed and reasons for discontinuing oral care, evaluated at the end of the study

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH de Brive, Brive-la-Gaillarde
  - CHU Limoges, Limoges

IPD SHARING:
Plan to Share IPD: No